CLINICAL TRIAL: NCT01461616
Title: Effect of NPH Insulin, Insulin Detemir and Insulin Glargine on IGFBP-1 Production and Serum IGF-I in Subjects With Type 1 Diabetes Mellitus: An Open-label, Randomised, Triple Cross-over Trial
Brief Title: Effect of NPH Insulin, Insulin Detemir and Insulin Glargine on GH-IGF-IGFBP Axis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NPH-Detemir-Glargine-2011
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Isophane Insulin, Human; Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NPH insulin injection (Experimental): NPH insulin will be injected in random order in one of three seperated visit days.
  Interventions: Drug: NPH
- detemir insulin injection (Experimental): insulin detemir will be injected in random order in one of three seperated visit days.
  Interventions: Drug: Detemir
- glargine insulin injection (Experimental): insulin glargine will be injected in random order in one of three seperated visit days.
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: NPH — equal doses of NPH insulin, insulin Detemir and insulin glargine injection
  Other Names: NPH insulin: Insulatard
  Arms: NPH insulin injection
Drug: Detemir — equal doses of NPH insulin, insulin Detemir and insulin glargine injection
  Other Names: insulin Detemir: Levemir
  Arms: detemir insulin injection
Drug: Glargine — equal doses of NPH insulin, insulin Detemir and insulin glargine injection
  Other Names: insulin glargine: Lamtus
  Arms: glargine insulin injection

SUMMARY:
The objective is to describe the interaction of equal doses of NPH insulin (Neutral Protamine Hagedorn), insulin Detemir and insulin glargine on IGFBP-1 (Insulin-like Growth Factor Binding Protein-1) production as well as immunoreactive and bioactive IGF-I (Insulin-like Growth Factor-I) after once-daily injection on three separate visits in type 1 diabetic subjects.

DETAILED DESCRIPTION:
Because of the importance of receptors activation and potential effects on the IGF system, a head-to-head comparison of the eventual differential impact of intermediate-acting human insulin (NPH), insulin detemir and insulin glargine on the growth hormone-insulin-like growth factor-insulin-like growth factor binding protein (GH-IGF-IGFBP) axis is relevant to be conducted for the safety assurance of insulin analogues. Therefore, this study aims to investigate whether the serum insulin profile obtained by once-daily injection of long-acting insulin analog, insulin detemir or insulin glargine, has a different impact on IGFBPs production and IGF-I concentrations (total IGF-I) bioactivity and tissue-availability as compared to that seen during treatment with intermediate-acting human insulin, NPH insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities.
2. Diagnosis of diabetes mellitus according to WHO criteria; history and clinical course consistent with type 1 diabetes mellitus.
3. Diagnosed with diabetes for more than 6 years and using continuous subcutaneous insulin infusion (CSII) at least 6 months at time of inclusion.
4. Total daily insulin dose between 0.4 and 1.4 units/kg (both values included)
5. HbA1c between 6% and 9% (both values included).
6. Age ≥ 18 years.
7. BMI between 18.5 and 28 kg /m2 (including both values).

Exclusion Criteria:

1. Known or suspected allergy to trial product(s) or related products.
2. Recurrent major hypoglycaemic episodes.
3. Heart: Unstable Angina Pectoris, AMI < 12 months or heart insufficiency classified according to NYHA III-IV
4. Blood Pressure: Severe uncontrolled hypertension with BP > 180/110 mmHg, sitting
5. Liver: Impaired hepatic function corresponding to serum-ALAT or basic phosphatase > 2 x upper reference limit of the local laboratory.
6. Kidneys: Impaired renal function corresponding to serum-creatinin > 150 μmol/l according to the local laboratory.
7. Any disease judged by the investigator to affect the trial.
8. Pregnancy, breast-feeding or the intention of becoming pregnant or fertile women not using adequate contraceptive measures - adequate contraceptive method is sterilisation, hysterectomy or current use of contraceptive pills or intra uterine device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
IGF-I(ng/ml) | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.
IGFBP-1(ng/ml) | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.
IGFBP-2(ng/ml) | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.
IGFBP-3(ng/ml) | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.
Growth Hormone(ng/ml) | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.

SECONDARY OUTCOMES:
plasma glucose concentration (mmol/L) after a single injection of either NPH insulin, insulin Detemir or insulin glargine | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.
insulin concentration (mmol/L) after a single injection of either NPH insulin, insulin Detemir or insulin glargine | 16 hours (from 18:00 to 10:00 next day)
  Hourly samples will be taken from 18:00 to 10:00 next day.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sandahl Christiansen, M.D., Principal Investigator — Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Thrailkill KM. Insulin-like growth factor-I in diabetes mellitus: its physiology, metabolic effects, and potential clinical utility. Diabetes Technol Ther. 2000 Spring;2(1):69-80. doi: 10.1089/152091599316775. PMID 11467325
- [Background] Bereket A, Lang CH, Wilson TA. Alterations in the growth hormone-insulin-like growth factor axis in insulin dependent diabetes mellitus. Horm Metab Res. 1999 Feb-Mar;31(2-3):172-81. doi: 10.1055/s-2007-978716. PMID 10226799
- [Background] Clemmons DR. Modifying IGF1 activity: an approach to treat endocrine disorders, atherosclerosis and cancer. Nat Rev Drug Discov. 2007 Oct;6(10):821-33. doi: 10.1038/nrd2359. PMID 17906644
- [Background] LeRoith D, Yakar S. Mechanisms of disease: metabolic effects of growth hormone and insulin-like growth factor 1. Nat Clin Pract Endocrinol Metab. 2007 Mar;3(3):302-10. doi: 10.1038/ncpendmet0427. PMID 17315038
- [Background] Brismar K, Fernqvist-Forbes E, Wahren J, Hall K. Effect of insulin on the hepatic production of insulin-like growth factor-binding protein-1 (IGFBP-1), IGFBP-3, and IGF-I in insulin-dependent diabetes. J Clin Endocrinol Metab. 1994 Sep;79(3):872-8. doi: 10.1210/jcem.79.3.7521354.
- [Background] Janssen JA, Jacobs ML, Derkx FH, Weber RF, van der Lely AJ, Lamberts SW. Free and total insulin-like growth factor I (IGF-I), IGF-binding protein-1 (IGFBP-1), and IGFBP-3 and their relationships to the presence of diabetic retinopathy and glomerular hyperfiltration in insulin-dependent diabetes mellitus. J Clin Endocrinol Metab. 1997 Sep;82(9):2809-15. doi: 10.1210/jcem.82.9.4180. PMID 9284701
- [Background] Hanaire-Broutin H, Sallerin-Caute B, Poncet MF, Tauber M, Bastide R, Rosenfeld R, Tauber JP. Insulin therapy and GH-IGF-I axis disorders in diabetes: impact of glycaemic control and hepatic insulinization. Diabetes Metab. 1996 Jul;22(4):245-50. PMID 8767170
- [Background] Ekman B, Nystrom F, Arnqvist HJ. Circulating IGF-I concentrations are low and not correlated to glycaemic control in adults with type 1 diabetes. Eur J Endocrinol. 2000 Oct;143(4):505-10. doi: 10.1530/eje.0.1430505. PMID 11022197
- [Background] Bolli GB, Owens DR. Insulin glargine. Lancet. 2000 Aug 5;356(9228):443-5. doi: 10.1016/S0140-6736(00)02546-0. No abstract available. PMID 10981882
- [Background] Hirsch IB. Insulin analogues. N Engl J Med. 2005 Jan 13;352(2):174-83. doi: 10.1056/NEJMra040832. No abstract available. PMID 15647580
- [Background] Heinemann L, Sinha K, Weyer C, Loftager M, Hirschberger S, Heise T. Time-action profile of the soluble, fatty acid acylated, long-acting insulin analogue NN304. Diabet Med. 1999 Apr;16(4):332-8. doi: 10.1046/j.1464-5491.1999.00081.x. PMID 10220208
- [Background] Kurtzhals P, Schaffer L, Sorensen A, Kristensen C, Jonassen I, Schmid C, Trub T. Correlations of receptor binding and metabolic and mitogenic potencies of insulin analogs designed for clinical use. Diabetes. 2000 Jun;49(6):999-1005. doi: 10.2337/diabetes.49.6.999. PMID 10866053
- [Background] Varewijck AJ, Goudzwaard JA, Brugts MP, Lamberts SW, Hofland LJ, Janssen JA. Insulin glargine is more potent in activating the human IGF-I receptor than human insulin and insulin detemir. Growth Horm IGF Res. 2010 Dec;20(6):427-31. doi: 10.1016/j.ghir.2010.10.002. Epub 2010 Nov 4. PMID 21055982
- [Background] Vigneri R, Squatrito S, Sciacca L. Insulin and its analogs: actions via insulin and IGF receptors. Acta Diabetol. 2010 Dec;47(4):271-8. doi: 10.1007/s00592-010-0215-3. Epub 2010 Aug 21. PMID 20730455
- [Background] Porcellati F, Rossetti P, Candeloro P, Lucidi P, Cioli P, Andreoli AM, Ghigo E, Bolli GB, Fanelli CG. Short-term effects of the long-acting insulin analog detemir and human insulin on plasma levels of insulin-like growth factor-I and its binding proteins in humans. J Clin Endocrinol Metab. 2009 Aug;94(8):3017-24. doi: 10.1210/jc.2008-2838. Epub 2009 May 26. PMID 19470629
- [Background] Slawik M, Schories M, Busse Grawitz A, Reincke M, Petersen KG. Treatment with insulin glargine does not suppress serum IGF-1. Diabet Med. 2006 Jul;23(7):814-7. doi: 10.1111/j.1464-5491.2006.01863.x. PMID 16842489